CLINICAL TRIAL: NCT04388150
Title: Efficacy of Narrow Band Spectrum Endoscopy Versus Histopathology for the Diagnosis of Gastric Antral Vascular Ectasia in Patients With Liver Cirrhosis
Brief Title: Efficacy of Narrow Band Spectrum Endoscopy for the Diagnosis of Gastric Antral Vascular Ectasia in Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Randa Salah, Assistant lecturer, Internal Medicine Department, Alexandria University
Other Study IDs: 0201288
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Gastric Antral Vascular Ectasia
Keywords: Narrow Band
MeSH Terms: conditions — Gastric Antral Vascular Ectasia | interventions — Endoscopy, Digestive System; Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Upper gastrointestinal endoscopy and biopsy — Gastroscope with technology of VIST video intelligent staining technology for taking biopsies

SUMMARY:
the study aims to evaluate the role of similar technology of Narrow Band Imaging VIST video intelligent staining technology in the diagnosis of Gastric Antral Vascular ectasia in cirrhotic patients

DETAILED DESCRIPTION:
VIST (Video intelligent staining technology) is used to the diagnosis of GAVE as the form of ectatic vessels in the antrum in instead of erosions in the antrum by White light endoscopy which can mislead the diagnosis to Portal hypertension gastropathy. Targeted biopsies are taken and examined histopathologically in order to see if matching with VIST view. In addition, CD61 is used to highlight the diagnosis for more confirmation. CD61 is an immunohistochemistry platelets marker.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mucosal vascular lesions at the gastric antrum suspicious of GAVE of a linear striped form or a diffuse punctate form upon conventional WLE

Exclusion Criteria:

* Connective tissue disorders like systemic sclerosis.
* Chronic kidney disease.
* Recent use of proton pump inhibitors in the last 14 days.
* History of gastric surgery or gastric cancer.
* Pernicious anemia.
* Recent history of non-steroidal anti-inflammatory drugs intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all cirrhotic patients undergoing Upper gastrointestinal endoscopy and they have antral erosions by endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Narrow Band Spectrum endoscopy for the diagnosis of Gastric antral vascular ectasia in cirrhotic patients | it is estimated to be 12 months
  It is done by the new technology of VIST which is similar to Narrow Band Imaging in the diagnosis of Gastric antral vascular ectasia in cirrhotic patients that were misdiagnosed before as portal hypertension gastropathy

CONTACTS AND LOCATIONS:
Overall Officials: Randa Salah Eldin Abdelmoneim, Master, Principal Investigator — Alexandria University
Locations (1):
- Internal Medicine, Hepatology Unit. Faculty of Medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided